CLINICAL TRIAL: NCT05940441
Title: A Prospective Exploratory Clinical Study of Metronomic Capecitabine as Adjuvant Therapy in Locoregionally Advanced Hypopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023060
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: to Explore Whether the Adjuvant Therapy of Metronomic Capecitabine Could Improve the Disease-free Survival of Locoregionally Advanced Hypopharyngeal Carcinoma
MeSH Terms: interventions — Capecitabine; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Capecitabine 500Mg Oral Tablet — 650 mg/m² body surface area twice daily for 1 year

SUMMARY:
To explore whether the adjuvant therapy of metronomic capecitabine could improve the disease-free survival of locoregionally advanced hypopharyngeal carcinoma (stage IV：T4N0-1M0，anyTN2-3M0).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 65 years old. 2. Histologically confirmed hypopharyngeal carcinoma, staged as IV (T4N0-1M0，anyTN2-3M0) (as defined by the 8th AJCC edition), Complete the recommended standard treatment (curative chemoradiotherapy, or radical surgery + postoperative chemo/radiotherapy ).

  3. No clinical evidence of persistent locoregional disease or distant metastases after definitive chemoradiotherapy.

  4. Within 8 weeks after completion of the last radiation dose. 5. Performance status of ECOG grade 0 or 1. 6. Adequate hematologic (neutrophil count > 1.5×10^9/L, hemoglobin > 90g/L and platelet count > 100×10^9 /L), hepatic (alanine aminotransferase, aspartate aminotransferase ≤ 1.5×ULN, bilirubin ≤ 1.5×ULN, alkaline phosphatase < 2.5×ULN) and renal function (creatinine clearance > 50 ml/min).

  7. Patients must be appraised of the investigational nature of the study and provide written informed consent.

Exclusion Criteria:

* 1.Patients who were known to be intolerable or allergic to capecitabine. 2. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.

  3. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control).

  4. With esophagus cancer. 5. Pregnancy or lactation. 6. Other conditions that are not eligible for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypopharyngeal carcinoma, staged as IV (T4N0-1M0，anyTN2-3M0) (as defined by the 8th AJCC edition), Complete the recommended standard treatment (curative chemoradiotherapy, or radical surgery + postoperative chemo/radiotherapy )
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2023.7-2025.7
  the time from enrolled to disease recurrence (distant metastasis or locoregional recurrence) or death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
the overall surviving results will be shared